CLINICAL TRIAL: NCT02670122
Title: Prospective, Multicenter, Non Randomized, Single Arm Study to Evaluate Safety of Transarterial Chemoembolization (TACE) With Doxorubicin Eluting 100 µ Microspheres in Patients With Non Resectable Hepatocellular Carcinoma
Brief Title: Prospective Study to Evaluate Safety of Deb-TACE With 100µ Beads in Patients With Non Resectable HCC
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, Jose Urbano Garcia, MD, PhD, EBIR, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Other Study IDs: FJD-TAN-14-01
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with non resectable HCC: DEB-TACE with doxorubicin eluting 100 µ microspheres
  Interventions: Device: DEB-TACE

INTERVENTIONS:
Device: DEB-TACE — Selective and ultraselective transcatheter intraarterial administration up to 3ml of well calibrated 100µ drug eluting microspheres with up to 150 mg of doxorubicin.

SUMMARY:
This is an observational, multicenter, single arm, prospective study to evaluate safety and tolerability of selective and ultraselective drug eluting beads transcatheter intraarterial chemoembolization (DEB-TACE) with up to 3 ml of well calibrated 100 µ microspheres and up to 150 mg of doxorubicin, for the treatment of non resectable hepatocellular carcinoma (HCC).

The hypothesis is that 100 µ beads penetrate deeper into the tumor than those eluting beads with larger volumes without increasing the risk and complications of DEB-TACE.

DETAILED DESCRIPTION:
In this observational, prospective study patients will undergo DEB-TACE and subsequent follow up procedures according to standard clinical practice. The primary aim of the study is to describe treatment safety and tolerability of 100 µ beads in DEB-TACE. As a secondary end-point a description of efficacy parameters will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of HCC according to European Association for the Study of the Liver (EASL) and American Association for the Study of Liver Diseases (AASLD) criteria and staged by BCLC criteria
2. Indication for receiving transarterial chemoembolization DEB-TACE with 100 µ microspheres according to usual clinical practice.
3. Able and willing to participate and give their written informed consent.
4. Both genders and ≥ 18 years old.
5. Eastern Cooperative Oncology Group (ECOG) 0
6. Preserved hepatic function (Child-Pugh ≤ B7).
7. No evidence of tumoral invasion in portal vein or main biliary ducts.
8. Able to go through image diagnostic techniques such as CT or MRI.
9. Preserved cardiac and renal function.
10. No concomitant active infections that require antibiotic treatment.
11. Measurable disease according to mRECIST criteria.
12. Life expectancy over 6 months.

Exclusion Criteria:

1. ECOG ≥ 1
2. Child-Pugh ≥B8.
3. Presence of ascitis or encephalopathy
4. Extrahepatic tumoral disease.
5. Tumoral vascular invasion
6. Serum bilirubin>3 mg/dl.
7. Cr Clearance ≤ 60 ml/min
8. If any of the following is contraindicated:

   1. Administration of doxorubicin
   2. Iodated contrasts
   3. CT or MRI procedures
   4. Transarterial embolization procedures
   5. White blood cells (WBC) < 2000 /mm3
   6. Neutrophil count < 1500 /mm3
   7. Ejection fraction < 50 %
   8. Platelet count < 5 x 104/mm3, international normalized ratio (INR) > 2,0)
   9. Transaminases (AST and/or ALT) > 5x upper limit of normal or >250 u/l
   10. Known hepatofugal portal vein flow
   11. A-V intrahepatic macroscopic fistula
9. Pregnant or breast feeding women.
10. Tumor burden involving more than 50% of the liver.
11. Active bacterial or fungal infection.
12. Other concomitant tumors.
13. Any other condition that according to investigator criteria, contraindicates DEB-TACE.
14. Patients not willing to participate and/or give their written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population includes:
  * Patients with stage B HCC carcinoma according to Barcelona Clinic Liver Cancer classification (BCLC).
  * Patients with stage A HCC according to BCLC if they are not candidates or not willing to go through surgery or radiofrecuency.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Urbano, MD, PhD,EBIR, Principal Investigator — HRyC
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Urbano J, Echevarria-Uraga JJ, Ciampi-Dopazo JJ, Sanchez-Corral JA, Cobos Alonso J, Anton-Ladislao A, Pena-Baranda B, Nacarino-Mejias V, Gonzalez-Costero R, Munoz Ruiz-Canela JJ, Perez-Cuesta J, Lanciego C, de Gregorio MA. Multicentre prospective study of drug-eluting bead chemoembolisation safety using tightly calibrated small microspheres in non-resectable hepatocellular carcinoma. Eur J Radiol. 2020 May;126:108966. doi: 10.1016/j.ejrad.2020.108966. Epub 2020 Mar 19. PMID 32278280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective inclusion from march 2015 to november 2016 in 10 University Hospitals
Period: Overall Study
Arm/Group | Patients With Non Resectable HCC
Started | 131
Completed | 127 (18 patients recieved liver transplantation)
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Non Resectable HCC
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.64 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 128
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 131
  Europe | 131
Technical success rate [Number; unit: DEB-TACE procedures] — Technical success is defined as the achievement of vascular stasis in the tumor feeding arteries or the administration of the full drug dose, with no technical complications during the DEB-TACE procedure.
  DEB-TACE procedures | 214

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Major and minor complications, procedure related mortality and post-embolisation syndrome after DEB-TACE of non-resectable HCC, using 100-µm doxorubicin-loaded microspheres
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Major Complications: Common Terminology Criteria for Adverse Events 4.03 grade 3 or 4 adverse events
- Minor Complications: Common Terminology Criteria for Adverse Events 4.03 grade 1 or 2 adverse events
- Procedure Related Mortality: Patients that died due to the DEB-TACE procedure
- Severe PES: Severe Post Embolisation Syndrome is when due to the pain and/or fever caused by the DEB TACE procedure requires intravenous analgesia and extend hospital admission.
Arm/Group | Major Complications | Minor Complications | Procedure Related Mortality | Severe PES
Number analyzed (Participants) | 131 | 131 | 131 | 131
Participants | 9 | 29 | 0 | 12

2. Secondary Outcome: Tumor Response
Description: Devascularization pattern in the treated tumor, assessed with the modified RECIST (mRECIST), in the contrast enhanced liver CT or MR obtained during FU.
Time Frame: 6 months, 1 year, 2 year
Measure: Count of Participants; unit: Participants
Groups:
- 6 m ORR: Objective Response Rate as the sum of complete and partial response rate 6 months after the first DEB-TACE
- 12 m ORR: Objective Response Rate as the sum of complete and partial response rate 12 months after the first DEB-TACE
- 24 m ORR: Objective Response Rate as the sum of complete and partial response rate 24 months after the first DEB-TACE
Arm/Group | 6 m ORR | 12 m ORR | 24 m ORR
Number analyzed (Participants) | 118 | 94 | 61
Participants | 90 | 42 | 27

3. Secondary Outcome: OS
Description: Overall survival
Time Frame: 2 years
Population: Patients that completed 2 year follow up. Patients losf for FU and the patients who recieved recieved liver transplantation are censored.
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- Overall Survival: OS is defined as the cumulative 24-month survival rate.
Arm/Group | Overall Survival
Number analyzed (Participants) | 109
months | 22 [13 to 24]

ADVERSE EVENTS:
Time Frame: 2 years
Description: CTCAE 4.03 criteria
Groups:
- Adverse Events: Mortality, minor and major adverse events after Tandem-100 DEB-TACE were assessed in accordance with CTCAE 4.03 criteria
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 48/131
Serious Adverse Events (participants affected / at risk) | 9/131
Other Adverse Events (participants affected / at risk) | 29/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=131)
Hepatic Abcess (Hepatobiliary disorders) | 3 (3)
Cholecistitis, conservative management (Hepatobiliary disorders) | 2 (2)
Worsening of a severe COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
HCC rupture and bleeding. Embolization 10h after TACE (General disorders) | 1 (1)
SIRS systemic inflammatory response syndrome, CKD chronic kidney disease. ICU (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=131)
Severe PES (General disorders) | 12 (12)
Asymptomatic segmentary bile duct/biliary tree dilatation (Hepatobiliary disorders) | 8 (8)
Asymtomatic segmental hepatic artery dissection (Vascular disorders) | 2 (2)
big groing hematoma (Vascular disorders) | 2 (2)
Biloma. Conservative treatment. (Hepatobiliary disorders) | 1 (1)
Asymptomatic coagulative thrombosis of a segmental portal branch (LWH) (Vascular disorders) | 1 (1)
Asymptomatic segmental hepatic artery perforation (Vascular disorders) | 1 (1)
Partial alopecia (General disorders) | 1 (1)
Periumbilical bruise (non target falciform artery embolization) (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
1. Lack of a comparative arm using larger or smaller DEBs or a cTACE group.
2. Intratumor doxorubicin doses were calculated according to the mL of injected mirospheres

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-03-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT02670122/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-03-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT02670122/Prot_SAP_001.pdf